CLINICAL TRIAL: NCT04490083
Title: Predictors of Pain Relief and Stone Fragmentation in Patients Undergoing Extra Corporeal Shock Wave Lithotripsy for Chronic Pancreatitis
Brief Title: Predictors of Pain Relief in Chronic Pancreatitis Undergoing ESWL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Sponsor
Other Study IDs: CP_ESWLPainrelief
Record Dates: First submitted 2020-07-21; First posted 2020-07-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Chronic Pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Extra corporeal shock wave lithotripsy — ESWL will be performed with a third generation electromagnetic lithotripter (Delta Compact, Dornier Med Tech, Germany) This has both fluoroscopy and ultrasound imaging facility. Radio opaque calculi will be targeted directly while a naso pancreatic tube (NPT) was placed for all radiolucent calculi and contrast was passed through this to localize the calculi. Between 5000 and 6000 shocks were delivered per session with frequency of 90 shocks per minute. The aim will be to fragment the calculi to <3 mm or demonstrate a decrease in heterogeneity or density of the calculi in the main pancreatic duct. Shocks will be delivered on consecutive days till fragmentation is achieved. If there is no fragmentation after four sessions of ESWL the procedure will be labeled as unsuccessful and patient will be advised surgery. Procedures will be performed under epidural anesthesia.

SUMMARY:
Extra corporeal shock wave therapy (ESWL) is recommended for pain management in patients with stone formation in pancreatic duct. ESWL can cause complete stone fragmentation and removal in 70% patients, associated with 85 to 90% pain relief.

Investigators aim to study, predictors pain relief in patients who undergo ESWL, to find out which patients will improve and which patients won't improve in terms of pain.

DETAILED DESCRIPTION:
The study will be a single center observational study.

General information of the patient in form of duration of symptoms and duration of diagnosis,exocrine and endocrine insufficiency. Imaging findings such as main pancreatic duct stone,size,parenchymal calcification , ductal stricture and its location, using any medications such as antioxidants and pain killers .

The pain score will be estimated by Izbicki's pain score in last 6 months. Patients will receive standard of care during study period, and they won't receive any experimental therapy.

After 6months of ESWL further general information of the patient any addictions, a formal imaging and determining main pancreatic duct stone ,size ,calcifications and strictures and also usage of any medications for decreasing pain.

Pain will be calculated by Izbick's pain score in last 6 months . Comparing pain score and information investigators will evaluate predictive factors of pain relief after ESWL by logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pancreatitis patients undergoing ESWL

Exclusion Criteria:

* Patients with multiple pancreatic duct stones
* Patients with multiple pancreatic duct strictures
* Pancreatic head mass
* Patients with ascites
* Pregnancy
* Patients not giving consent for participation
* Pseudocyst

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will be prospectively enrolled from patients with chronic pancreatitis undergoing ESWL in hospital.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients having persistent pain | 6 months
  Patients with persistent pain after 6 months of ESWL will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Jagtap, MD, DNB, Principal Investigator — Asian Institute of Gastroenterology, Hyderabad, India
Locations (1):
- Manu Tandan, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No